CLINICAL TRIAL: NCT03853733
Title: Palliative Hypofractionated Radiotherapy in Non-operable Rectal Cancer: A Retrospective Study
Brief Title: Hypofractionated Palliative Radiotherapy in Patients With Advanced Non-operable Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Joan Lozano Galan, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: ONCORTCST2019-2
Record Dates: First submitted 2019-02-18; First posted 2019-02-26 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
Keywords: palliative radiotherapy; rectal bleeding; hypofractionated radiotherapy
MeSH Terms: conditions — Rectal Neoplasms; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Radiation: rectal cancer radiotherapy — Conformal three-dimensional radiotherapy to deliver to the primary tumor and the enlarged pelvic nodes a total dose of 39Gy in 13 sessions of 3Gy in 17 days.

SUMMARY:
Many patients with rectal cancer were not candidates for surgical resection because advanced age, comorbidities, or multiple synchronous metastases. In this scenario only comfort measures or different palliative radiotherapy regimens are applied, from single doses to treatments lasting several weeks. The aim of this prospective study is to describe the preliminary results of our protocol of hypofractionated palliative radiotherapy in patients with non-operable rectal cancer.

DETAILED DESCRIPTION:
Many patients with rectal cancer were not candidates for surgical resection because advanced age, comorbidities, or multiple synchronous metastases. In this scenario only comfort measures or different palliative radiotherapy regimens are applied, from single doses to treatments lasting several weeks. The aim of this prospective study is to describe the preliminary results of our protocol of hypofractionated palliative radiotherapy in patients with non-operable rectal cancer.

Patients with rectal cancer who were not candidates for surgical resection because advanced age, comorbidities, or multiple synchronous metastases at the time of diagnosis were considered eligible.

Patients were immobilized in the prone position with a belly-board in order to reduce small bowel irradiation. To limit organ motion patient were instructed to empty the bladder and drink 500cm3 of water 45-60 minutes before CT simulation and before every treatment fraction.

A conformal three-dimensional radiotherapy technique was planned to deliver to the primary tumor and the enlarged pelvic nodes a total dose of 39Gy in 13 sessions of 3Gy in 17 days.

Symptomatic response after the end of treatment has been measured for bleeding and pain and acute toxicity were reported according to CTCAEv4.0 scale.

ELIGIBILITY:
Inclusion criteria :

1. Patients with rectal or sigmoidal cancer who were not candidates for surgical resection because advanced age, comorbidities, or multiple synchronous metastases at the time of diagnosis
2. Patients with = or > 18 years old
3. Patients treated with a radiotherapy dose of 39Gy in 13 fractions of 3 Gy

Exclusion criteria:

1. Patients with a non rectum or sigma colo-rectal cancer.
2. Patients with <18 years old.
3. Patients treated with concurrent chemotherapy
4. Patients candidates for surgical resection after radiotherapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer who were not candidates for surgical resection because advanced age, comorbidities, or multiple synchronous metastases at the time of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic response after palliative radiotherapy (bleeding) | two months afer the end of radiotherapy
  number of patients with bleeding ( worst, no change, better or without)
Symptomatic response after palliative radiotherapy (pain) | two months afer the end of radiotherapy
  number of patients with pain ( worst, no change, better or without)
Gastrointestinal toxicity after the end of radiotherapy | two months afer the end of radiotherapy
  Gastrointestinal toxicity after the end of radiotherapy were reported according to CTCAE v4.0 scale
Genitourinary toxicity after the end of radiotherapy | two months afer the end of radiotherapy
  Genitourinary toxicity after the end of radiotherapy were reported according to CTCAE v4.0 scale.

SECONDARY OUTCOMES:
palliative colostomy after the end of palliative radiotherapy | two months afer the end of radiotherapy
  number of patients with colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Joan Lozano, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] EP-1648: Palliative hipofractionated radiotherapy in non operable rectal cancer: preliminary results RSS Download PDF J. Lozano Galan, E. Rubio and J. Solé Radiotherapy and Oncology, 2018-04-01, Volume 127, Pages S887-S887